CLINICAL TRIAL: NCT06148038
Title: A Phase 1a "Window Trial" of Cannabidiol (CBD) For Breast Cancer Primary Tumors
Brief Title: CBD for Breast Cancer Primary Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 103565
Record Dates: First submitted 2023-04-17; First posted 2023-11-28 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a randomized placebo controlled double blind window of opportunity trial. A maximum of 120 patients will be enrolled. Up to 60 patients with invasive breast cancer will be enrolled into cohort 1, and up to 60 patients with DCIS will be enrolled into cohort 2. Patients in each cohort will be randomized 1:1 to either CBD or placebo control using permuted block randomization with random block sizes of 2 or 4. The time window between CBD or placebo initiation and surgery will be between 5 days and 56 days.
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CBD Oral (Experimental): CBD Oral 350mg twice daily for 28 days
  Interventions: Drug: CBD Oral
- Placebo control (Placebo Comparator): Placebo control Oral twice daily for 28 days
  Interventions: Other: Control

INTERVENTIONS:
Drug: CBD Oral — CBD Oral 350mg twice daily for 28 days
  Arms: CBD Oral
Other: Control — Placebo Control
  Arms: Placebo control

SUMMARY:
This is a randomized placebo controlled double blind window of opportunity trial. A maximum of 120 patients will be enrolled. Up to 60 patients with invasive breast cancer will be enrolled into cohort 1, and up to 60 patients with DCIS will be enrolled into cohort 2. Patients in each cohort will be randomized 1:1 to either CBD or placebo control using permuted block randomization with random block sizes of 2 or 4. The time window between CBD or placebo initiation and surgery will be between 5 days and 56 days.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed invasive breast cancer (stages I, II, or III) or DCIS with primary tumor(s) ≥ 0.8 cm on mammogram, ultrasound, MRI, or physical exam 2.18 years of age or older 3.Subject must understand risks and benefits of the protocol and be able to give informed consent 4.Women of child-bearing potential (WOCBP) must agree to use an approved form of birth control and to have a negative pregnancy test result before registration. WOCBP is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal. Menopause is defined clinically as 12 consecutive months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes.

5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 6.Adequate hematologic and end organ function, defined by the following laboratory results obtained within 14 days prior to registration:

* ANC ≥ 1.5 × 109/L
* Platelet count ≥ 100 × 109/L
* Hemoglobin ≥ 9 g/dL
* Albumin ≥ 2.5 g/dL
* Bilirubin ≤ 1.5 × the upper limit of normal (ULN)
* AST, ALT, and alkaline phosphatase ≤ 3 × ULN
* Serum creatinine ≤ 1.5 × ULN or creatinine clearance (CrCl) ≥ 40 mL/min on the basis of measured CrCl from a 24-hour urine collection or Cockcroft-Gault* glomerular filtration rate estimation:

  (140-age) × (weight in kg) × (0.85 if female) 72 × (serum creatinine in mg/dL)

  * The Modification of Diet in Renal Disease (Levey et al. 2006) and the Chronic Kidney Disease Epidemiology Collaboration (Levey et al. 2009) formulas for estimation of glomerular filtration rate are also acceptable.

  7. Ability and capacity to comply with the study and follow-up procedures 8. Subjects must be scheduled for surgery no less than 5 days from the planned start of day 1 and no more than 56 days from the planned start of day 1.

  9. If patients are taking home regimens of CBD or marijuana, they must consent to abstain for the length of the trial.

Exclusion Criteria:

1. Subjects undergoing neoadjuvant chemotherapy or neoadjuvant endocrine therapy
2. Subjects who are pregnant or are lactating.
3. Patients taking drugs metabolized by cytochrome p450 (warfarin, amiodarone, levothyroxine, clobazam, lamotrigine, valproate, prednisolone, hydrocortisone, clarithromycin, itraconazole, erythromycin, fluconazole, clopidogrel, rifampin, sulfamethoxazole, any opioids, antiepileptic medications (including carbamazapine, phenytoin, valproic acid, but excepting of gabapentin, clonazepam, or diazepam).
4. Routine use of recreational or medicinal marijuana products (defined as > 4 times per month) or illicit drug use including opioids, cocaine, amphetamines, PCP, LSD
5. Concurrent use of over-the-counter CBD oil, Marinol®, Delta-8 THC, or cannabis
6. History of allergic reactions attributed to compounds of similar chemical or biologic composition to CBD or placebo
7. Underlying history of epilepsy/ recurrent seizure disorder or unexplained seizure within past 6 months
8. Patients with uncontrolled cardiovascular disease defined by myocardial infarction, stroke, or transient ischemic attack, or need for coronary stent placement within past six months.
9. Patients with a psychiatric illness or psychiatric symptoms that would prevent them from completing study procedures or would disqualify them from surgical intervention (e.g., untreated schizophrenia, bipolar disorder, or suicide ideation/attempt resulting in psychiatric hospitalization within the last 30 days).
10. Women who are pregnant or breastfeeding or who refuse to practice an effective form of birth control (condoms, diaphragm, birth control pill, IUD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
CBD and cell proliferation | 2 months
  To determine whether oral administration of cannabidiol (CBD) causes biological changes related to cell proliferation (using Ki67 expression as a marker) in primary tumors of breast cancer patients.
CBD and apoptosis | 2 months
  To determine whether oral administration of cannabidiol (CBD) causes biological changes related to apoptosis (using Ki67 expression as a marker) in primary tumors of breast cancer patients.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE 5.0 | 2 months
  To determine adverse event relationship to oral CBD extract in patients with breast cancer.
GAD-7 anxiety level scoring at Pre and post CBD administration | 2 months
  To determine whether CBD administered in the period waiting for surgery reduces self-reported anxiety from baseline to time of surgery as measured by the GAD-7 patient reported outcomes scale.